CLINICAL TRIAL: NCT02797158
Title: Post TAVI Coronary REVASCularisation Guided by Myocardial Perfusion Imaging: a Prospective Open Label Pilot Study: The REVASC-TAVI Study
Acronym: REVASC-TAVI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RECHMPL15_0498; 2016-A00037-44 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2016-05-30; First posted 2016-06-13 (Estimated); Last update posted 2025-09-30 (Actual); Status verified 2019-05

CONDITIONS: Severe and Symptomatic Aortic Stenosis; Stable Coronary Disease
Keywords: TAVI; Aortic stenosis; Coronary artery disease; Coronary angiography; Percutaneous Coronary Intervention; Myocardial ischemia; SPECT; Coronary revascularization
MeSH Terms: conditions — Aortic Valve Stenosis; Coronary Artery Disease; Myocardial Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Interventional Arm (Experimental)
  Interventions: Procedure: TAVI procedure

INTERVENTIONS:
Procedure: TAVI procedure — Targeted and selected revascularization guided on myocardial ischemia detection after the TAVI procedure by using single photon emission computed tomography (SPECT) myocardial perfusion imaging.

SUMMARY:
Evaluation of a strategy of selected revascularization guided on myocardial ischemia detection after the TAVI procedure by using single photon emission computed tomography (SPECT) myocardial perfusion imaging.

DETAILED DESCRIPTION:
Background: Percutaneous coronary intervention (PCI) is usually proposed to patients with aortic stenosis (AS) before TransAortic Valve Implantation (TAVI) when significant coronary stenosis is detected on preprocedural coronary angiography. However, the benefit of a systematic revascularisation is unknown and may have specific complications in elderly and frail patients.

Aims: The investigators proposed a strategy of selected revascularization guided on myocardial ischemia detection after the TAVI procedure by using single photon emission computed tomography (SPECT) myocardial perfusion imaging.

Methods: This prospective open label clinical trial will include 71 consecutive patients with significant coronary artery disease (CAD) defined by one or more significant coronary stenosis in patients admitted for TAVI. Myocardial SPECT imaging will be performed in all patients at 1-month follow-up after the TAVI procedure. Targeted PCI will be performed only in patients with significant related ischemia (> 10 % myocardial perfusion defect).

The primary outcome criterion is a composite criterion of feasibility and safety including all causes of death, stroke, major bleedings, major vascular complications, per procedural myocardial infarction, coronary revascularization or rehospitalisation for cardiac cause at 6 month follow-up.

Hypothesis: An alternative management of CAD guided by significant myocardial ischemia detection after TAVI could reduce the risk of unnecessary revascularization, the complications and the costs inherent to these procedures and a phase II trial is requiring to the evaluate this innovative and less invasive strategy.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years
* Severe and symptomatic aortic stenosis defined as a median trans-valvular gradient higher than 40 mmHg and an aortic valve area of less than 1.0 cm2 or 0,6 cm2/m2 on echocardiography associated to significant CAD defined by ≥1 stenosis of ≥70% in a major epicardial coronary artery or ≥50% for left main
* Patients is not candidate for surgical aortic valve replacement after the multidisciplinary heart team decision.

Exclusion Criteria:

* Recent acute coronary syndrome (within 30 days before randomization),
* Unprotected left main disease
* Critical stenosis (>90%) of Left Anterior Descending artery (LAD),
* Significant angina (CCS class more than 2)
* Active bleeding,
* Contraindication for tomographic technetium-99 assessment or dipyridamole injection
* Previous enrollment in a other study
* Impossibly to obtain consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2016-06-23 (Actual); Primary Completion 2019-07-15 (Actual); Study Completion 2019-07-15 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is a composite of all cause of death | 6 months
  Mortality is defined as death due to any cause, the exact nature and date of which will be recorded. All deaths will be considered cardiovascular-related unless there is documentation to the contrary.
The primary endpoint is a composite of stroke | 6 months
The primary endpoint is a composite of major bleeding | 6 months
  Major bleedings are defined by ≥2 BARC classification.
The primary endpoint is a composite of major vascular complication | 6 months
  Access site complications is defined in accordance with the Valve Academic Research Consortium (VARC) guidelines.
The primary endpoint is a composite of periprocedural myocardial infarction | 6 months
  Perprocedural myocardial infarction is defined by 5-fold increased of basal troponin level associated to angina or ECG changes
The primary endpoint is a composite of hospitalization for cardiac cause. | 6 months

SECONDARY OUTCOMES:
Post-TAVI mortality | 1 and 6 months
Major adverse cardiovascular or cerebrovascular event (MACCE) | 1 and 6 months
Acute coronary syndrome (ACS) | 1 and 6 months
Acute myocardial infarction (MI) | 1 and 6 months
Rate of stroke | 1 and 6 months
Repeat revascularization by either PCI or CABG | 1 and 6 months
Hospitalization for heart failure or for non cardiovascular causes | 1 and 6 months
Duration of hospital stay | 1 and 6 months
Quality of life by Kansas city cardiomyopathy questionnaire | 1 and 6 months
Per-procedural complications | 1 and 6 months
  ventricular fibrillation (VF), ventricular tachycardia (VT) requiring cardioversion, cardiopulmonary arrest requiring cardiopulmonary resuscitation (CPR) and/or assisted mechanical respiratory support
percentage of pacemaker after implantation of the valve | 1 and 6 months
Bleeding complications according to the BARC classification | 1 and 6 months
Severe VARC Access Site Complications (Safety Issue at 1 and 6 months) | 1 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Florence LECLERCQ, PU PH, Principal Investigator — Montpellier University Hospital
Locations (1):
- Montpellier University Hospital, Montpellier, France

IPD SHARING:
Plan to Share IPD: No